CLINICAL TRIAL: NCT06360510
Title: Comparison of the Effectiveness of Ultrasound-guided 5% Dextrose and Betamethasone Injections in Patients With Carpal Tunnel Syndrome.
Brief Title: Comparison of %5 Dextrose and Betamethasone Injections in Patients With Carpal Tunnel Syndrome
Status: Active, not recruiting | Type: Observational
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Yasin Demir, MD, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: 44
Record Dates: First submitted 2024-04-07; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; betamethasone; % 5 dextrose
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Betamethasone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- %5 dextrose group
  Interventions: Procedure: %5 dextrose injection
- betamethasone group
  Interventions: Procedure: betamethasone injection

INTERVENTIONS:
Procedure: %5 dextrose injection — hydrodissection with %5 dextrose
  Groups: %5 dextrose group
Procedure: betamethasone injection — perineural betamethasone injection
  Groups: betamethasone group

SUMMARY:
The aim of the study is to compare the effectiveness of ultrasound-guided betamethasone and 5% dextrose injection, which is routinely applied in clinical practice, in patients with mild and moderate carpal tunnel syndrome (CTS).

DETAILED DESCRIPTION:
It is planned as an observational, single-center clinical study.A total of 28 patients diagnosed with mild-moderate carpal tunnel syndrome who meet the inclusion criteria will be included in the study.Patients who had been experiencing trigger finger symptoms for at least three month and who presented to the Gaziler Physical Medicine and Rehabilitation Training and Research Hospital, affiliated with the Health Sciences University Faculty of Medicine.

Patients will be divided into two groups. One group will receive 5% dextrose, the other group will receive 1 session of local injection by mixing Celeston chronodose [1ml/3 mg betamethasone acetate+3,947 mg betamethasone disodium phosphate (equivalent to 3 mg betamethasone)] and 1 ml 2% prilocaine.

Evaluations will be made before injection, at weeks 4 and 12.

ELIGIBILITY:
Inclusion Criteria:

* Paresthesia and pain symptoms in the region corresponding to the distribution of the median nerve
* Detection of mild or moderate CTS by electromyography
* One or both of the Phalen test and/or Tinel sign are positive on physical examination
* Symptoms have persisted for at least 3 months

Exclusion Criteria:

* Those diagnosed with polyneuropathy, plexopathy, radiculopathy, thoracic outlet syndrome
* Having had surgery or any injection for carpal tunnel syndrome within the last year
* History of wrist fracture
* Those with rheumatoid arthritis, uncontrolled diabetes, gout, chronic renal failure, malignancy, active systemic infection
* Those with cognitive impairment
* Coagulopathy or bleeding tendency
* Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients that have carpal tunnel syndrome
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2023-05-05 (Actual); Primary Completion 2024-05-05 (Estimated); Study Completion 2024-05-05 (Estimated)

PRIMARY OUTCOMES:
vas | three months

SECONDARY OUTCOMES:
boston carpal tunnel syndrome questionnaire | three months
median nerve cross sectional area | three months
tinnel test positivity | three months
phalen test positivity | three months
duruöz hand index | three months
global evaluation of treatment outcomes | three months

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Gaziler Physical Medicine and Rehabilitation Education and Research Hospital, Ankara, Turkey (Türkiye)